CLINICAL TRIAL: NCT02795780
Title: An Open Label, Multicenter Study Evaluating the Imaging Characteristics of a Follow up 18F-AV-1451 Scan in Subjects That Participated in the Confirmatory Cohort of 18F-AV-1451-A05
Brief Title: Follow up 18F-AV-1451 Scan in Confirmatory Cohort Subjects From Study 18F-AV-1451-A05
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A18
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Follow-up Flortaucipir PET Scan (Experimental)
  Interventions: Drug: Flortaucipir F18; Procedure: PET Scan

INTERVENTIONS:
Drug: Flortaucipir F18 — 370 megabecquerel (MBq) IV single-dose
  Other Names: T807; 18F-AV-1451
Procedure: PET Scan — positron emission tomography (PET) scan

SUMMARY:
This study will evaluate longitudinal change of tau deposition as measured by flortaucipir F 18 uptake over time.

ELIGIBILITY:
Inclusion Criteria:

* Confirmatory cohort subjects who completed the 18F-AV-1451-A05 (NCT02016560) study

Exclusion Criteria:

* Current clinically significant cardiovascular disease, ECG abnormalities, risk factors for Torsades de Pointes (TdP), or are taking drugs known to cause QT prolongation
* Current clinically significant infectious disease, endocrine or metabolic disease, pulmonary, renal or hepatic impairment, or cancer
* Females of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception
* Have had a non-study related radiopharmaceutical imaging or treatment procedure within 7 days prior to the study imaging session
* Have received or participated in a trial with investigational medications in the past 30 days

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Imaging Endpoints, Scottsdale, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Institute for Brain Aging and Dementia, UC Irvine, Irvine, California
  - 21st Century Oncology, Newport Beach, California
  - Alzheimer's Disease Center, UC Davis, Sacramento, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Compass Research, LLC, Orlando, Florida
  - Meridien Research, St. Petersburg, Florida
  - University of South Florida Health Byrd Alzheimer's Institute, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Las Vegas Radiology, Las Vegas, Nevada
  - New York University Center for Brain Health, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled between Aug 2016 and Aug 2017. The only subjects eligible were those who completed the Confirmatory Phase of Study A05 (NCT02016560).
Groups:
- AD Subjects: Clinically diagnosed dementia with a suspected neurodegenerative cause with an MMSE score ≥20 and ≤27
- MCI Subjects: Clinically diagnosed mild cognitive impairment with a suspected neurodegenerative cause with an MMSE score ≥20 and ≤27
Period: Overall Study
Arm/Group | AD Subjects | MCI Subjects
Started | 25 | 54
Completed | 25 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AD Subjects: Clinically diagnosed dementia with a suspected neurodegenerative cause with an MMSE score ≥20 and ≤27 from the flortaucipir PET scan arm
- MCI Subjects: Clinically diagnosed mild cognitive impairment with a suspected neurodegenerative cause with an MMSE score ≥20 and ≤27 from the flortaucipir PET scan arm
- Total: Total of all reporting groups
Arm/Group | AD Subjects | MCI Subjects | Total
Number analyzed (Participants) | 25 | 54 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.8 (10.63) | 73.2 (9.1) | 73.4 (9.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 22 | 31
  Male | 16 | 32 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 24 | 51 | 75
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 25 | 51 | 76
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 54 | 79
MMSE [Mean (Standard Deviation); unit: units on a scale] — Mini-mental status exam (MMSE) is a 30-point questionnaire that is used to measure cognitive impairment. Scores range from 0 to 30 with lower scores representing greater levels of cognitive impairment.
  units on a scale | 23.7 (2.39) | 25.9 (1.48) | 25.2 (2.06)
CDR-SB [Mean (Standard Deviation); unit: units on a scale] — The CDR scale (Berg 1988) examines 6 cognitive functioning domains individually on a scale of 0 to 3. CDR Sum of Boxes (CDR-SB) is generated by summing the total score across domains. Scores range from 0 to 18, with higher scores indicating higher levels of cognitive impairment.
  units on a scale | 4.8 (1.53) | 2.6 (1.91) | 3.3 (2.05)
Amyloid status [Count of Participants; unit: Participants] — Amyloid status (positive/negative) determined by florbetapir PET
  Participants
    Amyloid positive | 19 | 26 | 45
    Amyloid Negative | 6 | 28 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in Tau Deposition Over Time by Diagnostic Group and Amyloid Status
Description: Change in flortaucipir standardized uptake value ratio (SUVr) over 18 months. For SUVr, a value of 1 signifies no flortaucipir activity above background, values greater than 1 signify increasing flortaucipir activity in the brain. A positive change in SUVr represents an increase in tau deposition in the brain. Change = 18 month SUVr - baseline SUVr obtained in Study A05.
Time Frame: 18 months
Population: Excluded 1 MCI Aβ+ and 1 MCI Aβ- subject for whom 18 month follow-up clinical was not available
Measure: Least Squares Mean (Standard Deviation); unit: standardized uptake value ratio (SUVr)
Groups:
- AD Aβ+ Subjects: Amyloid positive AD subjects from the flortaucipir PET scan arm
- AD Aβ- Subjects: Amyloid negative AD subjects from the flortaucipir PET scan arm
- MCI Aβ+ Subjects: Amyloid positive MCI subjects from the flortaucipir PET scan arm
- MCI Aβ- Subjects: Amyloid negative MCI subjects from the flortaucipir PET scan arm
Arm/Group | AD Aβ+ Subjects | AD Aβ- Subjects | MCI Aβ+ Subjects | MCI Aβ- Subjects
Number analyzed (Participants) | 19 | 6 | 26 | 26
standardized uptake value ratio (SUVr) | 0.0205 (0.01871) | -0.0912 (0.03619) | 0.0352 (0.01185) | -0.0124 (0.01185)
Statistical Analysis 1: Comparison: AD Aβ+ Subjects vs AD Aβ- Subjects; Test of whether difference in least squares mean change is 0; Test type: Other; p = 0.0166, ANCOVA — No adjustments for multiplicity. No a priori threshold defined; Adjusted for baseline SUVr, age, and diagnosis group (AD/MCI)
Statistical Analysis 2: Comparison: MCI Aβ+ Subjects vs MCI Aβ- Subjects; Test of whether difference in least squares mean change is 0; Test type: Other; p = 0.0108, ANCOVA — No adjustments for multiplicity. No a priori threshold defined; Adjusted for baseline SUVr, age, and diagnosis group (AD/MCI)

ADVERSE EVENTS:
Time Frame: 48 hours after study drug administration
Description: Adverse events (AEs) were collected at scan visits, regardless of attribution to study drug. AEs occurring after study drug administration, but outside that window were not recorded, unless considered attributable to study drug.
Groups:
- MCI Subjects: MCI subjects receiving a dose of flortaucipir
- AD Subjects: AD subjects receiving a dose of flortaucipir
Arm/Group | MCI Subjects | AD Subjects
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/25
Other Adverse Events (participants affected / at risk) | 2/54 | 0/25
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MCI Subjects (N=54) | AD Subjects (N=25)
injection site pain (General disorders) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
flushing (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-03-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT02795780/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT02795780/SAP_001.pdf